CLINICAL TRIAL: NCT03212638
Title: A Bioequivalence and Food Effect Study in Healthy Subjects Comparing Baricitinib Suspension and Commercial Tablet Formulations
Brief Title: A Study of Baricitinib in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 14934; I4V-MC-JAGU (Other: Eli Lilly and Company)
Record Dates: First submitted 2017-07-07; First posted 2017-07-11 (Actual); Results first posted 2019-03-26 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Healthy
MeSH Terms: interventions — baricitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Baricitinib T1 (Part A) (Experimental): 4 mg (milligram) baricitinib suspension test formulation (TF) administered orally (PO) without water following a 10 hour fast. (Baricitinib T1)
  Interventions: Drug: Baricitinib suspension
- Baricitinib T2 (Part A) (Experimental): 4 mg baricitinib suspension formulation (TF) administered PO prior to 240 mL water following a 10 hour fast (Baricitinib T2)
  Interventions: Drug: Baricitinib suspension
- Baricitinib R (Part A) (Experimental): 4 mg baricitinib tablet administered PO, taken with 240 mL water following a 10 hour fast (baricitinib R)
  Interventions: Drug: Baricitinib tablet
- Baricitinib TF Fasted (Part B) (Experimental): 4 mg baricitinib suspension test formulation (TF) administered after 10 hour fast. (TF fasting)
  Interventions: Drug: Baricitinib suspension
- Baricitinib TF Fed (Part B) (Experimental): 4 mg baricitinib suspension TF administered after a high fat meal.(baricitinib TF Fed)
  Interventions: Drug: Baricitinib suspension

INTERVENTIONS:
Drug: Baricitinib suspension — Administered orally
  Other Names: LY3009104
  Arms: Baricitinib T1 (Part A); Baricitinib T2 (Part A); Baricitinib TF Fasted (Part B); Baricitinib TF Fed (Part B)
Drug: Baricitinib tablet — Administered orally
  Other Names: LY3009104
  Arms: Baricitinib R (Part A)

SUMMARY:
The purposes of this study are to determine:

* If there are any differences in the amount of baricitinib in the blood/body when taken in two different forms.
* How a high-fat, high-calorie meal affects the amount of baricitinib in the blood/body.
* The safety and tolerability of baricitinib.

The study has two parts. Individuals will participate in only one part.

Participants will be admitted to the clinical research unit (CRU) and will be discharged from the CRU following the completion of 3 overnight stays.

Each part of this study will last from 8-10 days, not including screening. Follow-up will occur 7 to 14 days after the last dose of baricitinib.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy males or females, as determined by medical history and physical examination
* Women not of child-bearing potential
* Have a body mass index (BMI) of 18.5 to 29.9 kilograms per meter squared (kg/m²) inclusive, at screening

Exclusion Criteria:

* Have received live vaccine(s) within 3 months of screening, or intend to during the study
* Have a current or recent history (less than [<] 30 days prior to screening and/or <45 days prior to Day -1 in Period 1) of a clinically significant bacterial, fungal parasitic, viral (not including rhinopharyngitis), or mycobacterial infection

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Singapore, Singapore

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A: Sequence ABC: A: 4 mg baricitinib suspension administered orally (PO) without water following a 10 hour fast. (Baricitinib T1)
  B: 4 mg baricitinib suspension administered PO prior to 240 mL water following a 10 hour fast (Baricitinib T2)
  C: 4 mg baricitinib tablet administered PO, taken with 240 mL water following a 10 hour fast (baricitinib R)
  With a 72 hour washout between doses
- Part A: Sequence BCA: B: 4 mg baricitinib suspension administered PO prior to 240 mL water following a 10 hour fast (Baricitinib T2)
  C: 4 mg baricitinib tablet administered PO, taken with 240 mL water following a 10 hour fast (baricitinib R)
  A: 4 mg baricitinib suspension administered orally (PO) without water following a 10 hour fast. (Baricitinib T1)
  With a 72 hour washout between doses
- Part A: Sequence CAB: C: 4 mg baricitinib tablet administered PO, taken with 240 mL water following a 10 hour fast (baricitinib R)
  A: 4 mg baricitinib suspension administered orally (PO) without water following a 10 hour fast. (Baricitinib T1)
  B: 4 mg baricitinib suspension administered PO prior to 240 mL water following a 10 hour fast (Baricitinib T2)
  With a 72 hour washout between doses
- Part B: Sequence DE: D: 4 mg baricitinib suspension test formulation (TF) administered when fasting (TF fasting).
  E:4 mg baricitinib suspension TF administered after a high fat meal.(baricitinib TF Fed)
  With a 72 hour washout between doses
- Part B:Sequence ED: E: 4 mg baricitinib suspension TF administered after a high fat meal.(baricitinib TF Fed)
  D: 4 mg baricitinib suspension test formulation (TF) administered when fasting. (TF fasting)
  With a 72 hour washout between doses
Period: Period 1
Arm/Group | Part A: Sequence ABC | Part A: Sequence BCA | Part A: Sequence CAB | Part B: Sequence DE | Part B:Sequence ED
Started | 8 | 8 | 8 | 0 | 0
Received at Least 1 Dose of Study Drug | 8 | 8 | 8 | 0 | 0
Completed | 8 | 8 | 8 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Part A: Sequence ABC | Part A: Sequence BCA | Part A: Sequence CAB | Part B: Sequence DE | Part B:Sequence ED
Started | 8 | 8 | 8 | 0 | 0
Received at Least 1 Dose of Study Drug | 8 | 8 | 8 | 0 | 0
Completed | 8 | 8 | 8 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Part A: Sequence ABC | Part A: Sequence BCA | Part A: Sequence CAB | Part B: Sequence DE | Part B:Sequence ED
Started | 8 | 8 | 8 | 0 | 0
Received at Least 1 Dose of Study Drug | 8 | 8 | 8 | 0 | 0
Completed | 8 | 8 | 8 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | Part A: Sequence ABC | Part A: Sequence BCA | Part A: Sequence CAB | Part B: Sequence DE | Part B:Sequence ED
Started | 0 (Participants were not allowed to participate in Part B and have completed study.) | 0 (Participants were not allowed to participate in Part B and have completed study.) | 0 (Participants were not allowed to participate in Part B and have completed study.) | 9 (New Participants in Part B, no participants from Part A participated in Part B.) | 9 (New Participants in Part B, no participants from Part A participated in Part B.)
Received at Least 1 Dose of Study Drug | 0 | 0 | 0 | 9 | 9
Completed | 0 | 0 | 0 | 9 | 9
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Period 5
Arm/Group | Part A: Sequence ABC | Part A: Sequence BCA | Part A: Sequence CAB | Part B: Sequence DE | Part B:Sequence ED
Started | 0 | 0 | 0 | 9 | 9
Received at Least 1 Dose of Study Drug | 0 | 0 | 0 | 9 | 9
Completed | 0 | 0 | 0 | 9 | 9
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants in Part A or Part B that received at least 1 dose of study drug.
Groups:
- Part A:All Participants: All participants who received study drug during Part A.
- Part B: All Participants: All participants who received study drug during Part B.
- Total: Total of all reporting groups
Arm/Group | Part A:All Participants | Part B: All Participants | Total
Number analyzed (Participants) | 24 | 18 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.9 (8.5) | 41.1 (11.3) | 40.4 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 23 | 18 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 24 | 18 | 42
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 24 | 17 | 41
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Singapore | 24 | 18 | 42
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per meter squared (kg/m^2)] | 24.14 (2.55) | 25.36 (3.03) | 24.5 (2.8)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of Baricitinib Following a Single Oral Dose
Description: PK: Cmax of baricitinib after a single oral dose
Time Frame: Predose, 0.25 hour (hr), 0.5 hr, 0.75 hr, 1 hr, 1.5 hr, 2 hr, 3 hr, 4 hr, 6 hr, 9 hr, 12 hr, 24 hr, 36 hr, 48 hr postdose
Population: All participants who received at least 1 dose of study drug and had evaluable PK parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Groups:
- Part A: Baricitinib T1: 4 mg baricitinib suspension administered orally (PO) without water following a 10 hour fast. (Baricitinib T1)
- Part A: Baricitinib T2: 4 mg baricitinib suspension administered PO prior to 240 mL water following a 10 hour fast (Baricitinib T2)
- Part A: Baricitinib R: 4 mg baricitinib tablet administered PO, taken with 240 mL water following a 10 hour fast (baricitinib R)
- Part B: Baricitinib TF Fasted: 4 mg baricitinib suspension test formulation (TF) administered after 10 hour fast (TF fasting).
- Part B: Baricitinib TF Fed: 4 mg baricitinib suspension TF administered after a high fat meal.(baricitinib TF Fed)
Arm/Group | Part A: Baricitinib T1 | Part A: Baricitinib T2 | Part A: Baricitinib R | Part B: Baricitinib TF Fasted | Part B: Baricitinib TF Fed
Number analyzed (Participants) | 24 | 24 | 24 | 17 | 18
nanograms per milliliter (ng/mL) | 49.8 (21) | 49.6 (24) | 47.8 (25) | 47.9 (22) | 32.5 (22)
Statistical Analysis 1: Comparison: Part A: Baricitinib T1 vs Part A: Baricitinib R; Bioequivalence of single 4 mg dose of baricitinib as the suspension formulation with (T1) water compared to the commercial tablet (R); Test type: Equivalence — 0.80, 1.25 as the bioequivalence boundaries; Ratio = 1.04, 95% CI 2-sided [0.946 to 1.15]
Statistical Analysis 2: Comparison: Part A: Baricitinib T2 vs Part A: Baricitinib R; Bioequivalence of single 4 mg dose of baricitinib as the suspension formulation without (T2) water compared to the commercial tablet (R); Test type: Equivalence — 0.80, 1.25 as the bioequivalence boundaries; ratio = 1.04, 95% CI 2-sided [0.944 to 1.14]
Statistical Analysis 3: Comparison: Part B: Baricitinib TF Fasted vs Part B: Baricitinib TF Fed; Bioequivalence of single 4 mg dose of baricitinib as fasted vs fed; Test type: Equivalence — 0.80, 1.25 as the bioequivalence boundaries; Ratio = 0.675, 95% CI 2-sided [0.617 to 0.740]

2. Primary Outcome: PK: Area Under the Concentration Versus Time Curve From Time Zero to the Last Time Point With a Measurable Concentration (AUC[0-tlast]) of Baricitinib Following a Single Oral Dose
Description: PK: AUC(0-tlast) of Baricitinib, measured in hour times nanogram per milliliter (ng*hr/mL)
Time Frame: as for outcome 1
Population: All participants who received at least 1 dose of study drug and had evaluable PK parameters.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Part A: Baricitinib T1 | Part A: Baricitinib T2 | Part A: Baricitinib R | Part B: Baricitinib TF Fasted | Part B: Baricitinib TF Fed
Number analyzed (Participants) | 24 | 24 | 24 | 17 | 18
ng*hr/mL | 314 (19) | 315 (17) | 216 (18) | 281 (22) | 273 (20)
Statistical Analysis 1: Comparison: Part A: Baricitinib T1 vs Part A: Baricitinib R; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — 0.80, 1.25 as the bioequivalence boundaries; Ratio = 0.996, 95% CI 2-sided [0.963 to 1.03]
Statistical Analysis 2: Comparison: Part A: Baricitinib T2 vs Part A: Baricitinib R; Bioequivalence of s single 4 mg dose of baricitinib as the suspension formulation without (T2) water compared to the commercial tablet (R); Test type: Equivalence — 0.80, 1.25 as the bioequivalence boundaries; Ratio = 0.998, 95% CI 2-sided [0.995 to 1.03]
Statistical Analysis 3: Comparison: Part B: Baricitinib TF Fasted vs Part B: Baricitinib TF Fed; Bioequivalence of single 4 mg dose of baricitinib as fasted vs fed; Test type: Equivalence — 0.80, 1.25 as the bioequivalence boundaries; ratio = 0.973, 95% CI 2-sided [0.936 to 1.01]

3. Primary Outcome: PK: Area Under the Concentration Versus Time Curve From Time Zero to Infinity (AUC[0-∞]) of Baricitinib Following a Single Oral Dose
Description: PK: AUC(0-∞) of Baricitinib
Time Frame: as for outcome 1
Population: All participants who received at least 1 dose of study drug and had evaluable PK parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Part A: Baricitinib T1 | Part A: Baricitinib T2 | Part A: Baricitinib R | Part B: Baricitinib TF Fasted | Part B: Baricitinib TF Fed
Number analyzed (Participants) | 24 | 24 | 24 | 17 | 18
ng*hr/mL | 319 (19) | 319 (17) | 319 (17) | 284 (22) | 282 (21)
Statistical Analysis 1: Comparison: Part A: Baricitinib T1 vs Part A: Baricitinib R; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — 0.80, 1.25 as the bioequivalence boundaries; Ratio = 0.999, 95% CI 2-sided [0.996 to 1.03]
Statistical Analysis 2: Comparison: Part A: Baricitinib T2 vs Part A: Baricitinib R; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — 0.80, 1.25 as the bioequivalence boundaries; Ratio = 0.999, 95% CI 2-sided [0.966 to 1.03]
Statistical Analysis 3: Comparison: Part B: Baricitinib TF Fasted vs Part B: Baricitinib TF Fed; Bioequivalence of single 4 mg dose of baricitinib as fasted vs fed; Test type: Equivalence — 0.80, 1.25 as the bioequivalence boundaries; ratio = 0.978, 95% CI 2-sided [0.941 to 1.02]

ADVERSE EVENTS:
Time Frame: Baseline through end of study (Up to 120 days)
Arm/Group | Part A: Baricitinib T1 | Part A: Baricitinib T2 | Part A: Baricitinib R | Part B: Baricitinib TF Fasted | Part B: Baricitinib TF Fed
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 2/24 | 1/24 | 4/24 | 1/18 | 5/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Baricitinib T1 (N=24) | Part A: Baricitinib T2 (N=24) | Part A: Baricitinib R (N=24) | Part B: Baricitinib TF Fasted (N=18) | Part B: Baricitinib TF Fed (N=18)
Catheter site bruise (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Catheter site pain (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site swelling (General disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-09-28): https://cdn.clinicaltrials.gov/large-docs/38/NCT03212638/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-05): https://cdn.clinicaltrials.gov/large-docs/38/NCT03212638/SAP_001.pdf